CLINICAL TRIAL: NCT06702241
Title: Neonatal Hyperbilirubinemia - Phototherapeutic Treatment Strategies
Brief Title: Newborn Jaundice - An Investigation of Different Approaches to Light Therapy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240019; F2024-032 (Other: The North Denmark Region)
Record Dates: First submitted 2024-11-06; First posted 2024-11-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Cycled phototherapy; high irradiance phototherapy; Neonatal jaundice; Newborn jaundice; neonatal hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: All infants will receive 12 hours double therapy with a biliblanket and overhead light providing an intensity of either 40-, 55- or 70 µW/cm2/nm. Three groups will be treated with continuous phototherapy while a fourth group will receive intermittent phototherapy of 1,5 hours cycled intervals with an intensity of 70 µW/cm2/nm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 12 hours continuous double phototherapy with irradiance of over head light of 40 µW/cm2/nm (Active Comparator)
  Interventions: Other: Continuous Phototherapy with a irradiance of 40 µW/cm2/nm from the overhead light
- 12 hours continuous double phototherapy with irradiance of over head light of 55 µW/cm2/nm (Active Comparator)
  Interventions: Other: Continuos Phototherapy with a irradiance of 55 µW/cm2/nm from the overhead light
- 12 hours continuous double phototherapy with irradiance of over head light of 70 µW/cm2/nm (Active Comparator)
  Interventions: Other: Continuous Phototherapy with a irradiance of 70 µW/cm2/nm from the overhead light
- 12 hours cycled double phototherapy with irradiance of over head light of 70 µW/cm2/nm (Active Comparator): This group will receive 12 hours double phototherapy in cycles of 1,5 hours. Thus receiving 1,5 hours treatment, 1,5 hours pause, 1,5 hours treatment etc.
  Interventions: Other: Cycled phototherapy with a irradiance of 70 µW/cm2/nm from the overhead light

INTERVENTIONS:
Other: Continuous Phototherapy with a irradiance of 40 µW/cm2/nm from the overhead light — The difference in irradiance between the groups will be measured with a radiometer specific to the device's wavelength.
  Arms: 12 hours continuous double phototherapy with irradiance of over head light of 40 µW/cm2/nm
Other: Continuos Phototherapy with a irradiance of 55 µW/cm2/nm from the overhead light — The difference in irradiance between the groups will be measured with a radiometer specific for the device's wavelenght
  Arms: 12 hours continuous double phototherapy with irradiance of over head light of 55 µW/cm2/nm
Other: Continuous Phototherapy with a irradiance of 70 µW/cm2/nm from the overhead light — The difference in irradiance between the groups will be measured with a radiometer specific for the device's wavelenght
  Arms: 12 hours continuous double phototherapy with irradiance of over head light of 70 µW/cm2/nm
Other: Cycled phototherapy with a irradiance of 70 µW/cm2/nm from the overhead light — The difference in irradiance between the groups will be measured with a radiometer specific for the device's wavelenght
  Arms: 12 hours cycled double phototherapy with irradiance of over head light of 70 µW/cm2/nm

SUMMARY:
Background Neonatal jaundice affects about 60% of full-term newborns in their first week. If untreated, it can lead to permanent brain damage. In Denmark, 2-5% of newborns require phototherapy, the standard treatment. The maximum beneficial irradiance limit for phototherapy remains unclear. Furthermore, studies suggest that cycled phototherapy is as effective as continuous treatment.

This study aims to investigate the efficacy of elevating the irradiance of intensive phototherapy treatment regimens. This is to evaluate the dose-response relationship. Furthermore, the study aims to compare intermittent phototherapy to continuous phototherapy.

Methods:

In a clinical randomized multicenter trial 116 newborns with non-hemolytic hyperbilirubinemia, gestational age >33+0, weight >1800g and no other significant neonatal diagnose will be randomized. All infants will receive 12 hours double therapy with a biliblanket and overhead light providing an intensity of either 40-, 55- or 70 µW/cm2/nm. Three groups will be treated with continuous phototherapy while a fourth group will receive intermittent phototherapy of 1,5 hours cycled intervals with an intensity of 70 µW/cm2/nm.

Parental experiences during treatment will be examined through a survey post treatment.

The study has been approved by the Regional Research Ethics Committee.

Perspectives:

Understanding the dose-response relationship of phototherapy will give an insight in the most effective way of treating neonatal jaundice. Intermittent therapy, if proven non-inferior, could facilitate more intimacy in the parent-infant relationship as well as benefits in initiating breastfeeding

DETAILED DESCRIPTION:
A randomized clinical study is planned to determine whether there is an upper limit to the efficacy of phototherapy irradiance and whether intermittent/cyclic treatment is as effective as continuous treatment. The study will be conducted at the Maternity Ward and the Department of Pediatrics and Adolescents at the North Denmark Regional Hospital, as well as the Neonatal Department at Aalborg University Hospital. Power calculations require the inclusion of 29 children in each of the four groups, totaling 116 children.

Inclusion criteria are newborns born at ≥33+0 weeks of gestation and a birth weight of ≥1800 g, with a blood bilirubin level above the treatment threshold as specified in the national guidelines. Newborns with rapidly rising bilirubin levels, indicating the need for more intensive treatment with light from multiple sides, exchange transfusion, or possibly immunoglobulin, are excluded from the study.

All children will be treated with double light-overhead light and a light blanket-for 12 hours. The included children will be randomized into one of four groups, each with a specific irradiance level for overhead phototherapy: 40, 55, and 70 µW/cm²/nm. The light blanket under the child will provide an irradiance of 30 µW/cm²/nm. The 70 µW/cm²/nm group will be divided into two subgroups: continuous and intermittent treatment. Thus, there will be four groups in total. Irradiance can be measured and practically adjusted by modifying the distance between the child and the light source. For intermittent treatment, a strategy of 1.5 hours of phototherapy followed by a 1.5-hour pause will be used, based on experiences from other studies and to accommodate the family's and child's feeding needs.

The primary outcome is the reduction in total serum bilirubin, measured from the start of treatment to after 12 hours. Secondary outcomes will include recording whether any children experience a rebound increase in bilirubin. This will be done by reviewing the medical records of the included children to determine if a new blood test for serum bilirubin has been performed, indicating a rebound.

The children will be closely monitored for signs of early bilirubin encephalopathy through medical examinations, weight control, and records of food intake (either breast milk or formula). Serum bilirubin will be measured before the start of treatment. After 12 hours of treatment, serum bilirubin, hemoglobin, and photoisomers will be measured. Serum bilirubin must be measured no more than three hours before the start of phototherapy.

Data analysis will examine:

Differences between the three groups with varying light intensities. Differences between the two groups with the same irradiance but differing treatment regimens (intermittent vs. continuous).

Parents of children meeting the inclusion criteria will be presented with the project verbally and in writing by department staff in a quiet, undisturbed setting. Parents will have time to consider the project while awaiting blood test results and preparing for phototherapy. If parents cannot agree or decide, the child will not participate in the project.

The project is registered with the Research Projects Registry of the North Denmark Region (ID: F2024-032). The project is approved by the Danish Scientific Ethical Committee for Region North Jutland, registration number N-20240019.

Perspectives The study aims to enable more effective and shorter treatment for the 2-5% of all newborns receiving phototherapy. This will allow for more time to establish breastfeeding and bonding between the child and parent.

ELIGIBILITY:
Inclusion Criteria:

* Hyperbilirubinemia with a total serum bilirubin level above the limit of necessary treatment according to the Danish Pediatric Society's guidelines
* Birth weight >1800g
* Gestational age >33+0

Exclusion Criteria:

* Hyperbilirubinemia within the first 24 hours of life
* Rapidly increasing serum levels of bilirubnemia indicating pathology or hemolysis

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Total serum bilirubin | At 12 hours from initiated treatment

SECONDARY OUTCOMES:
Re-admissions to the hospital | 14 days after initiation of treatment the patient's file will be examined to determine, if relapse of the conidition has occured
Breast feeding or formula | At the initiation and immediately after treatment, as well as during a follow-up telephone call 4 months later.
  A description of the newborn's nutrition will be noted comparing cycled and continuous phototherapy. This is relevant because in continuous (standard) treatment the infant spends longer periods away from the parent thus making the establishment of breast feeding more difficult

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, The Neonatal Department, Aalborg
  - The North Denmark Regional Hospital, The Pediatric Department, Hjørring

IPD SHARING:
Plan to Share IPD: No
It is stated in the approval from the ethical comittee that no person outsite the project might gain knowledge or insight in IPD